CLINICAL TRIAL: NCT02900443
Title: A Randomised, Open-label Clinical Trial Assessing the Efficacy and Safety of Mycophenolate Mofetil Versus Azathioprine for Induction of Remission in Treatment Naive Autoimmune Hepatitis
Brief Title: Mycophenolate Mofetil Versus Azathioprine in Treatment Naive Autoimmune Hepatitis
Acronym: CAMARO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL57115.058.16
Record Dates: First submitted 2016-08-17; First posted 2016-09-14 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2021-10

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate mofetil (Experimental): The intervention group will receive oral mycophenolate mofetil for 24 weeks. Both groups will be treated with steroid induction which will closely follow the schedule from the recent EASL Clinical Practice Guidelines.
  Interventions: Drug: Mycophenolate mofetil
- Azathioprine (Active Comparator): . The control group will be treated with azathioprine (standard of care) for 24 weeks. Both groups will be treated with steroid induction which will closely follow the schedule from the recent EASL Clinical Practice Guidelines.
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Mycophenolate mofetil
  Arms: Mycophenolate mofetil
Drug: Azathioprine
  Arms: Azathioprine

SUMMARY:
Rationale: Current standard therapy of autoimmune hepatitis consists of a combination of prednisolone and azathioprine. However, a significant proportion of patients does not respond to, or is intolerant for, azathioprine. Mycophenolate mofetil (MMF) has surpassed azathioprine as therapy to prevent organ transplant rejection and is sometimes used as an alternative option for autoimmune hepatitis. Several case series and one prospective study have documented the efficacy and safety of mycophenolate mofetil as induction therapy for autoimmune hepatitis. Robust evidence from a formal randomized clinical trial is lacking.

Objective: To assess the efficacy and safety of mycophenolate mofetil as induction therapy in patients with treatment naive autoimmune hepatitis.

Study design: Multicenter, randomised, open-label intervention study Study population: Patients with newly diagnosed autoimmune hepatitis who are in need of induction therapy according to current guidelines.

Intervention: The intervention group will receive oral mycophenolate mofetil for 24 weeks. The control group will be treated with azathioprine for 24 weeks. Both groups will be treated with steroid induction which will closely follow the schedule from the recent Clinical Practice Guidelines by the European Association for Study of the Liver (EASL).

Main study parameters/endpoints: The primary outcome is the proportion of patients in biochemical remission, defined as normalization of serum alanine transaminase (ALT) and immunoglobulin G (IgG) levels after 24 weeks of treatment, per treatment group. Secondary endpoints include safety and tolerability of mycophenolate mofetil, time to remission, changes in Model For End-Stage Liver Disease (MELD) -score (and its components bilirubin, INR, creatinine), albumin, pseudocholinesterase and N-terminal procollagen-III-peptide, ELF (Enhanced Liver Fibrosis) -score and aspects of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Probable or definite diagnosis of autoimmune hepatitis according to the International Autoimmune Hepatitis Study Group criteria
* First presentation of AIH requiring treatment according to the current EASL guidelines
* Age ≥ 18 years
* Must provide informed consent and agree to comply with the trial protocol

Exclusion Criteria:

* Overlap syndrome with Primary Sclerosing Cholangitis (PSC) or Primary Biliary Cholangitis (PBC) (Paris criteria, strong positive Anti-Mitochondrial Antibodies (AMA), past liver biopsy or cholangiographic findings compatible with PBC or PSC).
* Presentation with acute liver failure, defined as presence of hepatic encephalopathy and coagulopathy (INR > 1.5)
* Current treatment with prednisone/prednisolone and/or immunosuppressive medication for an indication other than autoimmune hepatitis
* Current systemic infection
* Other clinically significant medical conditions that could interfere with the trial
* If female of childbearing potential: known pregnancy, or unwilling to practice anticontraceptive measures.
* History of noncompliance with medical regimens, or patients who are considered to be potentially unreliable or unable to participate
* Mental instability or incompetence, such that the validity of informed consent or compliance with the trial is uncertain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-01; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission | 24 weeks
  The percentage of patients in biochemical remission, defined as normalization of serum ALT and IgG levels after 24 weeks of treatment, per treatment group.

SECONDARY OUTCOMES:
Time to biochemical remission | 24 weeks
Biochemical remission at any time | Up to 24 weeks
Complete biochemical response, defined as normalization of AST, ALT and IgG at 6 months after initiation of treatment | Up to 24 weeks
Insufficient response, defined as lack of complete biochemical response determined at 6 months | Up to 24 weeks
Non-response at 4 weeks: defined as <50% decrease of serum transaminases within 4 weeks after initiation of treatment | Up to 4 weeks
Changes in MELD score (and its components bilirubin, international normalized ratio (INR), creatinine) and in albumin | Up to 24 weeks
Changes in liver stiffness, measured by transient elastography | Up to 24 weeks
N-terminal procollagen-III-peptide, ELF score | 24 weeks
Changes in quality of life measured with SF-36 | Up to 24 weeks
Difference in side-effects, adverse events and serious adverse events | Up to 24 weeks
The level of ALT, AST, GGT in both groups | Up to 24 weeks
Percentage of patients with biochemical remission | Up to 24 weeks
Ratio of ALT to lowest ALT ever | Up to 24 weeks
Extrahepatic AIH manifestations (e.g. arthralgia) | Up to 24 weeks
Patient survival | Up to 24 weeks
Fatigue index | Up to 24 weeks
Pruritis VAS score | Up to 24 weeks
Difference in cumulative corticosteroid dose between MMF and azathioprine | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Hoek, MD, PhD, Principal Investigator — Leiden University Medical Center; Joost PH Drenth, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (14):
- University Hospital Antwerpen, Antwerp, Belgium
- Netherlands (13):
  - Zuyderland, Heerlen, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Amsterdam UMC, location AMC, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Maastricht UMC+, Maastricht
  - Sint Antonius Hospital, Nieuwegein
  - Radboud University Medical Centre, Nijmegen
  - Erasmus MC, Rotterdam
  - Bernhoven, Uden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Snijders RJALM, Stoelinga AEC, Gevers TJG, Pape S, Biewenga M, Tushuizen ME, Verdonk RC, de Jonge HJM, Vrolijk JM, Bakker SF, Vanwolleghem T, de Boer YS, Baven Pronk MAMC, Beuers U, van der Meer AJ, Gerven NMFV, Sijtsma MGM, van Eijck BC, van IJzendoorn MC, van Herwaarden M, van den Brand FF, Korkmaz KS, van den Berg AP, Guichelaar MMJ, Levens AD, van Hoek B, Drenth JPH; Dutch Autoimmune Hepatitis Working Group. An open-label randomised-controlled trial of azathioprine vs. mycophenolate mofetil for the induction of remission in treatment-naive autoimmune hepatitis. J Hepatol. 2024 Apr;80(4):576-585. doi: 10.1016/j.jhep.2023.11.032. Epub 2023 Dec 14. PMID 38101756